CLINICAL TRIAL: NCT06285617
Title: Short-Term Versus 6-Week Prednisone in The Treatment of Subacute Thyroiditis: An Open-label, Randomized, Controlled, and Multicenter Trial
Brief Title: Short-Term Versus 6-Week Prednisone in The Treatment of Subacute Thyroiditis
Acronym: SAT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Lian Duan, Clinical Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022GDRC016
Record Dates: First submitted 2024-01-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Subacute Thyroiditis
Keywords: Short-Term Prednisone; Subacute Thyroiditis; Open-label, Randomized, Controlled, and Multicenter
MeSH Terms: conditions — Thyroiditis, Subacute

STUDY DESIGN:
Intervention Model Description: Prednisone
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group received 20 and 10 mg prednisone in the morning and afternoon, respectively, daily for 1 week; in the second week, these participants received 400 mg celecoxib on Day 1 and 200 mg twice daily for the remaining 6 days until celecoxib withdrawal.
  Interventions: Drug: 1-week predisone+1-week celecoxib
- Control group (Active Comparator): Participants in the control group received 20 and 10 mg prednisone in the morning and afternoon, respectively, daily in the first week, and then reduced by 5 mg/week from the second week until withdrawal in the sixth week.
  Interventions: Drug: 6-weeks predisone

INTERVENTIONS:
Drug: 1-week predisone+1-week celecoxib — 20 and 10 mg prednisone in the morning and afternoon, respectively, daily for 1 week; in the second week, these participants received 400 mg celecoxib (a type of nonsteroidal anti-inflammatory drug) on day 1 and 200 mg twice daily for the remaining 6 days until celecoxib withdrawal.
  Other Names: No available
  Arms: Experimental group
Drug: 6-weeks predisone — 20 and 10 mg prednisone in the morning and afternoon, respectively, daily in the first week, and then reduced by 5 mg/week from the second week until withdrawal in the sixth week.
  Other Names: No available
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of short-term versus 6-week prednisone in the treatment of moderate-to-severe subacute thyroiditis. The main questions it aims to answer are: Does the short-term medication regimen reduce glucocorticoid side effects while achieving similar efficacy as the guideline treatment group? Patients with moderate-to-severe symptoms were randomly assigned to receive either 30 mg/day prednisone for 1 week, followed by 1 week of nonsteroidal anti-inflammatory drugs, or the conventional 6-week prednisone therapy in the control group.

DETAILED DESCRIPTION:
This is an open-label, randomized, controlled, and multicenter trial. Patients with moderate-to-severe symptoms were randomly assigned to receive either 20 and 10 mg prednisone in the morning and afternoon, respectively, daily for 1 week; in the second week, these participants received 400 mg celecoxib on day 1 and 200 mg twice daily for the remaining 6 days until celecoxib withdrawal or 20 and 10 mg prednisone in the morning and afternoon, respectively, daily in the first week, and then reduced by 5 mg/week from the second week until withdrawal in the sixth week. The primary endpoint was intergroup differences in treatment efficacy at the end of the treatment course. Secondary endpoints included between-group differences in post-withdrawal adverse effect parameters and thyroid function at weeks 6, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled adult patients (age 18-70) with Subacute Thyroiditis (SAT) scores ≥3 points. SAT was diagnosed on the basis of diagnostic criteria. The severity of SAT was scored as follows: fever - none, <38℃, and >38℃ (0, 1, and 2 points, respectively); tenderness - none, mild, and severe (0, 1, and 2 points, respectively); goiter by ultrasonography or palpation - none and yes (0 and 1 point, respectively); and ESR - normal, 25-60 mm/h, and >60 mm/h (0, 1, and 2 points, respectively).

Exclusion Criteria:

* Patients who were diagnosed with diabetes, an active peptic ulcer, benign and malignant tumors, hepatic dysfunction, recurrent SAT, and already on glucocorticoid therapy were excluded within 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The difference in efficacy between the two groups at the completion. | The palpation and CRP will investigate at 2nd (experimental group) or 6th (control group) weeks.
  Efficacy is defined as no pain in the thyroid region through palpation and pain assessment using visual analog scoring, and normalization of CRP level.

SECONDARY OUTCOMES:
Thyroid function | Thyroid function will be measured at weeks 6, 12, and 24 after the initial treatment.
  The differences in thyroid function (FT3, FT4, TSH) between the two groups at the end of treatment.
Total cholesterol (TC) | TC will be measured at 2nd (experimental group) or 6th (control group) weeks.
  The differences in TC between the two groups at the end of treatment.
Triglycerides (TG) | TG will be measured at 2nd (experimental group) or 6th (control group) weeks.
  The differences in TG between the two groups at the end of treatment.
Systolic blood pressure (SBP) | SBP will be measured at 2nd (experimental group) or 6th (control group) weeks.
  The differences in SBP between the two groups at the end of treatment.
Diastolic blood pressure (DBP) | DBP will be measured at 2nd (experimental group) or 6th (control group) weeks.
  The differences in DBP between the two groups at the end of treatment.
Parathyroid hormone (PTH) | PTH will be measured at 2nd (experimental group) or 6th (control group) weeks.
  The differences in PTH between the two groups at the end of treatment.

REFERENCES:
- [Background] Duan L, Feng X, Zhang R, Tan X, Xiang X, Shen R, Zheng H. Short-Term Versus 6-Week Prednisone In The Treatment Of Subacute Thyroiditis: A Randomized Controlled Trial. Endocr Pract. 2020 Aug;26(8):900-908. doi: 10.4158/EP-2020-0096. PMID 33471681
- [Background] Alves C, Robazzi TC, Mendonca M. Withdrawal from glucocorticosteroid therapy: clinical practice recommendations. J Pediatr (Rio J). 2008 May-Jun;84(3):192-202. doi: 10.2223/JPED.1773. PMID 18535733
- [Background] Benbassat CA, Olchovsky D, Tsvetov G, Shimon I. Subacute thyroiditis: clinical characteristics and treatment outcome in fifty-six consecutive patients diagnosed between 1999 and 2005. J Endocrinol Invest. 2007 Sep;30(8):631-5. doi: 10.1007/BF03347442. PMID 17923793
- [Background] Kubota S, Nishihara E, Kudo T, Ito M, Amino N, Miyauchi A. Initial treatment with 15 mg of prednisolone daily is sufficient for most patients with subacute thyroiditis in Japan. Thyroid. 2013 Mar;23(3):269-72. doi: 10.1089/thy.2012.0459. PMID 23227861
- [Background] Waljee AK, Rogers MA, Lin P, Singal AG, Stein JD, Marks RM, Ayanian JZ, Nallamothu BK. Short term use of oral corticosteroids and related harms among adults in the United States: population based cohort study. BMJ. 2017 Apr 12;357:j1415. doi: 10.1136/bmj.j1415. PMID 28404617
- [Background] Broersen LH, Pereira AM, Jorgensen JO, Dekkers OM. Adrenal Insufficiency in Corticosteroids Use: Systematic Review and Meta-Analysis. J Clin Endocrinol Metab. 2015 Jun;100(6):2171-80. doi: 10.1210/jc.2015-1218. Epub 2015 Apr 6. PMID 25844620
- [Background] Oray M, Abu Samra K, Ebrahimiadib N, Meese H, Foster CS. Long-term side effects of glucocorticoids. Expert Opin Drug Saf. 2016;15(4):457-65. doi: 10.1517/14740338.2016.1140743. Epub 2016 Feb 6. PMID 26789102
- [Background] Pearce EN, Farwell AP, Braverman LE. Thyroiditis. N Engl J Med. 2003 Jun 26;348(26):2646-55. doi: 10.1056/NEJMra021194. No abstract available. PMID 12826640
- See also: This is the published small sample, single center, randomized controlled studies. Short-Term Versus 6-Week Prednisone In The Treatment Of Subacute Thyroiditis: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/33471681/